CLINICAL TRIAL: NCT03569423
Title: Comparison Between TPRK Versus AAPRK in Correction of Myopia and Myopic Astigmatism
Brief Title: Comparison Between TPRK Versus AAPRK in Correction of Myopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Hossam Mohamed Moharram, Assistant professor of ophthalmology, Minia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MiniaU2
Record Dates: First submitted 2018-04-27; First posted 2018-06-26 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Refractive Surgery; Myopia
MeSH Terms: conditions — Myopia | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: Prospective, consecutive, nonrandomized case-control comparative study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transepithelial PRK (Experimental): Transepithelial photorefractive keratectomy was done in 100 right eyes of 100 patients included in the study.
  Interventions: Procedure: Transepithelial photorefractive keratectomy; Procedure: Alcohol assisted photorefractive keratectomy
- Alcohol assisted PRK (Active Comparator): Alcohol assisted photorefractive keratectomy was done in 100 left eyes of the same 100 patients included in the study.
  Interventions: Procedure: Transepithelial photorefractive keratectomy; Procedure: Alcohol assisted photorefractive keratectomy

INTERVENTIONS:
Procedure: Transepithelial photorefractive keratectomy — ablations were performed with the Schwind Amaris excimer LASER 750S. Paired student's t-tests and Mann-Whitney tests were used for statistical analysis.
  Other Names: TPRK
Procedure: Alcohol assisted photorefractive keratectomy — ablations were performed with the Schwind Amaris excimer LASER 750S. Paired student's t-tests and Mann-Whitney tests were used for statistical analysis.
  Other Names: APRK

SUMMARY:
PURPOSE: The aim of the study is to compare visual acuity means, refractive results, safety, and efficacy of TPRK with AAPRK as primary outcomes and surgical time, pain scores, haze levels, and healing time as secondary outcomes.

SETTING: Security Forces Hospital, Ophthalmology Department, Riyadh, Kingdom of Saudi Arabia.

DESIGN: Prospective, consecutive, nonrandomized case-control comparative study.

. METHODS: A total of 200 eyes of 100 patients were included. One hundred eyes underwent TPRK in the right eye (study group) and 100 eyes underwent AAPRK in the left eye (control group). Ablations performed with the Schwind Amaris, 750S. Clinical outcomes were compared Paired student's t-tests and Mann-Whitney tests were used for statistical analysis.

DETAILED DESCRIPTION:
Introduction Previous studies document that, although Laser in situ keratomileusis (LASIK) is the most worldwide performed refractive procedure, surface ablation may be safer to avoid flap complications, corneal weakening, and a higher risk of iatrogenic keratectasia associated with LASIK and thus the era of surface ablation emerged as an alternative (1). Photorefractive keratectomy (PRK) is one of the surface ablation procedures and performed after corneal epithelial debridement accompanied by post-operative pain, discomfort, and high grade of corneal haze, all of which limit its popularity (2). The traditional method for corneal epithelium removal before excimer LASER was manual scraping, which was later enhanced by using an alcohol solution 20% or brush (3). In 2003, Camellin introduced a new alcohol-assisted technique called laser-assisted subepithelial keratectomy (LASEK) that allowed the epithelium to be preserved as a flap and applied back to the stromal corneal bed after laser treatment (4). Also in 2003, Pallikaris invented epithelial laser in situ keratomileusis (Epi-LASIK) which is another method that uses the epithelial flap and performed with a microkeratome (called epi-keratome) with a blunt oscillating blade. After trans-epithelial photorefractive keratectomy (TPRK) was introduced, where removal of the epithelium is done by phototherapeutic ablation followed by refractive ablation of the corneal stroma. Several studies emerged and advocated many techniques for epithelial removal , but this 2-step technique was not worldwide used due to the prolonged surgery time with the older generation of lasers, corneal dehydration, increased post-operative pain, and a deficiency of adjusted nomograms (5). When new generations of faster lasers, improved ablation algorithms, and nomograms have emerged, it allowed development of a new TPRK non touch: all-surface ablation technique which allows ablation the corneal epithelium and stroma in a single-step with one ablation profile. This aspheric profile is calculated according to data from the literature estimating that the normal corneal epithelial thickness is 55 μm centrally and 65 peripherally at 4 mm radially from the center (6). A number of recent studies demonstrated that this single-step TPRK is a relatively new procedure with many advantages such as, reduced surgical time, minimizing the size of epithelial defect to that required for stromal ablation, no alcohol use avoiding potential toxicity to the limbal cells, less post-operative pain and corneal haze with rapid healing time and faster visual recovery (7).Thus, there is a need for an updated comparative evaluation based on a larger number of eyes. The aim of our study is to compare 6-months un-corrected distant visual acuity (UDVA) and best corrected distant visual acuity (BCDVA) means, refractive results, safety, and efficacy of single-step TPRK with alcohol-assisted PRK (AAPRK) as primary outcomes and comparison of surgical time, pain scores, and haze levels, complete epithelial healing time, as secondary outcomes among the two procedures when used to correct mild to moderate myopia and myopic astigmatism.

Subjects and methods This study is a prospective, consecutive, nonrandomized case-control study that includes eyes that underwent either single-step TPRK or AAPRK between February 2017 and April 2018, at the Security Forces Hospital, Ophthalmology department, Riyadh, Kingdom of Saudi Arabia. The study was approved by the local ethical board committee. Before the surgical procedure, each patient was adequately informed about the study as well as the risks and benefits of the surgery, and signed informed consent in accordance with the Declaration of Helsinki.

A total of 200 eyes of 100 consecutive patients were included; One hundred eyes underwent TPRK (study group) and 100 eyes underwent AAPRK (control group). The study design choice of the procedure was fixed for each patient: the right eye underwent TPRK and the contra-lateral left eye AAPRK. Patients demographics and preoperative variables are demonstrated in Table (1). There are no significant differences in pre-operative variables of patients in the TPRK and AAPRK groups except the patients' genders. The percentage of females is 77% and males 23%. Patients who attended all visits, without any missing data, were included in the statistical analysis.

Preoperative Examination The preoperative examination included UDVA, BCDVA, manifest and cycloplegic refraction, slit lamp biomicroscopy, tonometry, Pentacam camera (OCULUS- Netzteil Art., pentacam HR, Germany), tomography (Sirius, SCHWIND eye-tech-solutions GmbH, Kleinostheim, Germany), and dilated fundus examination using binocular ophthalmoscopy. Contact lenses use and medical history, including any systemic diseases, were recorded.

Surgical Technique All surgeries were performed with 6th-generation Amaris excimer LASER 193, version 750 S (Schwind eye-tech-solutions GmbH& Co.KG, Mainparkstrasse, Kleinostheim, Germany). Ablations were based on aberration-free algorithms calculated using ORK-CAM software with beam size 0.54 mm full width and high-speed eye tracking. Treatments were performed by 2 surgeons (BA & ESH ) using an identical surgical protocol. The treatments were mostly aimed at emmetropia. Before the surgery, tetracaine hydrochloride 0.5% ophthalmic solution (Bausch & Lomb, Minims) and moxifloxacin 0.5% (Vigamox, Alcon Co.) drops were instilled 3 times within a 5-minutes interval. The eyelids were prepared with antiseptic Chlorohexidine Gluconate 0.05% solution (Saudi Medical Solution Company) and opened using a wire lid speculum. In the AAPRK group, the cornea was exposed to a 20% ethyl alcohol solution for 25 seconds with the use of a well. Subsequently, a superficial cut of the epithelium was made with either an 8.5 or 9.5 mm diameter trephine. The epithelium was mechanically debrided with the well or with a blunt spatula, then LASER treatment with the same machine was initiated. In the TPRK group, where aspheric aberration-free TPRK ablation algorithm was used (Schwind eye-tech-solutions), the epithelium was removed during laser ablation only from the area of the total ablation zone. In both groups and in all cases, immediately after treatment, the eye was washed with a balanced salt solution (BSS) for 20 seconds. Then, to fight against post-operative corneal haze, mitomycin C 0.02% (MMC) was applied for 30 seconds followed by copious irrigation of the eye with BSS. Intra-operative complications were not noted and surgical time starting from eye lid speculum insertion to the time of its removal at the end of the procedure were recorded. After the surgery, a bandage contact lens was applied (BIOMEDICS Evolution CL ocufilcon D 45%, water 55%) for 7 days. The postoperative regimen included tobradex eye drops 0.3% (Tobramycin 0.3% - dexamethazone 0.1% sterile eye drops, Alcon Co.) with tapering dose for 1 month starting with QID/ 1 week, TID/ 1 week, BID/ 1 week and once a day/1 week, moxifloxacin drops 0.5% (Vigamox, Alcon Co.) for 2 weeks, and sodium hyaluronate 0.2% (Hyfresh eye drops, Jamjoom Pharma Co.) drop / 2 hours and a gradual decreasing of the frequency for 3 months. Pain killer oral medication tablet/ 6 hours was used in the first post-operative days if needed.

Postoperative Examinations Patients were instructed to visit the clinic for postoperative examinations and follow up after 1 day, 1 week, 1 month, 3 months and 6 months. Examinations at 1 day, 1 week, 1 month, 3 months, and 6 months included UDVA ,but the BCDVA and manifest refraction were measured at 1, 3, and 6 months. Slit lamp biomicroscopy was done in each visit. Corneal haze grading was evaluated according to Fantes et al., 1990 proposal (0 = no haze; 0.5 = trace haze on oblique illumination; 1 = corneal cloudiness not interfering with the visibility of fine iris details; 2 = mild effacement of fine iris details; 3 and 4 = details of the lens and iris not discernible). Healing time in which complete re-epithelialisation occurred in both eyes were recorded. In post-operative day 1, day 3 and week 1, We used a discrete, 11-category numeric pain scale (NPS, 0 = no pain and 10 = the worst possible pain) to evaluate pain score in each eye and patients response were recorded at early postoperative period. Six months post-operatively, patients were asked about the overall satisfaction with each procedure as high, moderate, low, and not satisfied, and whether they would decide to have the surgery again (yes, no) were recorded.

Statistical Analysis Patients' data were entered in Microsoft Excel, copied and analyzed using Sigma Plot-Scientific Data Program for the 2 groups, Paired student's t-test was used for the UDVA & BCDVA means in decimal values and for MRSE means. Mann-Whitney test was used for pain scores, haze levels, and healing time. For all tests, a (P value < 0.05) was considered statistically significant. A Graph Pad Prism 5 program was used for graphs constructions.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Primary myopia or compound myopic astigmatism
* Preoperative manifest refraction spherical equivalent (MRSE) within the range of -1.50 to -7 D
* Stable refraction for at least 1 year before the surgery
* Contact lens discontinuation for at least 3 weeks
* Estimated stromal corneal bed thickness of >330 μm at the thinnest location.

Exclusion Criteria:

* Previous ocular surgery
* Active ocular diseases
* Corneal dystrophy
* Retinal disease
* Glaucoma
* Dry eye
* History of severe eye trauma
* Irregular astigmatism or suspected keratoconus on corneal topography
* Systemic disease that could affect corneal wound healing such as collagen diseases, diabetes mellitus, and pregnancy.

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2018-04-15 (Actual); Study Completion 2018-04-25 (Actual)

PRIMARY OUTCOMES:
Visual acuity means | 6 months
  visual acuity means in decimal value from minimum 0.1 to maximum 1.2.

SECONDARY OUTCOMES:
Surgical time | 6 months
  surgical time in seconds
Pain scores | 6 months
  pain scores,from 0 -10, 11-category numeric pain scale (NPS, 0 = no pain and 10 = the worst possible pain)
Haze levels | 6 months
  haze levels from 0 o 4 (0 = no haze; 0.5 = trace haze on oblique illumination; 1 = corneal
Complete epithelial healing time | 6 months
  complete epithelial healing time in days.

CONTACTS AND LOCATIONS:
Overall Officials: Shaaban A Elwan, MD, Principal Investigator — Minia University
Locations (2):
- Shaaban A Elwan, Al Minyā, Egypt
- Security forces hospital, Riyadh, Central, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Leaming DV. Practice styles and preferences of ASCRS members--2003 survey. J Cataract Refract Surg. 2004 Apr;30(4):892-900. doi: 10.1016/j.jcrs.2004.02.064. PMID 15093657
- [Result] Blake CR, Cervantes-Castaneda RA, Macias-Rodriguez Y, Anzoulatous G, Anderson R, Chayet AS. Comparison of postoperative pain in patients following photorefractive keratectomy versus advanced surface ablation. J Cataract Refract Surg. 2005 Jul;31(7):1314-9. doi: 10.1016/j.jcrs.2004.11.046. PMID 16105600
- [Result] Abad JC, An B, Power WJ, Foster CS, Azar DT, Talamo JH. A prospective evaluation of alcohol-assisted versus mechanical epithelial removal before photorefractive keratectomy. Ophthalmology. 1997 Oct;104(10):1566-74; discussion 1574-5. doi: 10.1016/s0161-6420(97)30095-5. PMID 9331192
- [Result] Camellin M. Laser epithelial keratomileusis for myopia. J Refract Surg. 2003 Nov-Dec;19(6):666-70. doi: 10.3928/1081-597X-20031101-09. PMID 14640432
- [Result] Carr JD, Patel R, Hersh PS. Management of late corneal haze following photorefractive keratectomy. J Refract Surg. 1995 May-Jun;11(3 Suppl):S309-13. doi: 10.3928/1081-597X-19950502-25. PMID 7553113
- [Result] Sin S, Simpson TL. The repeatability of corneal and corneal epithelial thickness measurements using optical coherence tomography. Optom Vis Sci. 2006 Jun;83(6):360-5. doi: 10.1097/01.opx.0000221388.26031.23. PMID 16772894
- [Result] Fadlallah A, Fahed D, Khalil K, Dunia I, Menassa J, El Rami H, Chlela E, Fahed S. Transepithelial photorefractive keratectomy: clinical results. J Cataract Refract Surg. 2011 Oct;37(10):1852-7. doi: 10.1016/j.jcrs.2011.04.029. Epub 2011 Aug 15. PMID 21840678
- [Derived] Bakhsh AM, Elwan SAM, Chaudhry AA, El-Atris TM, Al-Howish TM. Comparison between Transepithelial Photorefractive Keratectomy versus Alcohol-Assisted Photorefractive Keratectomy in Correction of Myopia and Myopic Astigmatism. J Ophthalmol. 2018 Nov 12;2018:5376235. doi: 10.1155/2018/5376235. eCollection 2018. PMID 30538854